CLINICAL TRIAL: NCT01387828
Title: Prospective Randomized Comparison of Open Versus Laparoscopic Management of Splenic Artery Aneurysms. A Ten-Year Study
Brief Title: Comparison Between Open and Laparoscopic Splenic Aneurysms Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Guido A M Tiberio, MD, AOBrescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOB 01-11
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-06

CONDITIONS: Splenic Artery Aneurysm
Keywords: Splenic artery; Aneurysm; laparoscopic; Vascular reconstruction; Splenectomy
MeSH Terms: conditions — Aneurysm | interventions — Splenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopy (Active Comparator): Includes all patient underwent intervention with a laparoscopic approach, even if converted to open surgery during intervention
  Interventions: Procedure: Laparoscopic splenic aneurysm repair, eventual splenectomy
- Open surgery (Active Comparator): Includes all the patients underwent intervention with a laparotomic approach; it does not include patient underwent laparoscopic approach and then converted in laparotomy.
  Interventions: Procedure: Laparotomic splenic artery aneurysm repair, eventual artery reconstruction or splenectomy

INTERVENTIONS:
Procedure: Laparoscopic splenic aneurysm repair, eventual splenectomy — Aneurysmectomy and eventual artery reconstruction or splenectomy performed with a laparoscopic approach
  Arms: Laparoscopy
Procedure: Laparotomic splenic artery aneurysm repair, eventual artery reconstruction or splenectomy — Aneurysmectomy and eventual artery reconstruction or splenectomy performed with a laparotomic approach
  Arms: Open surgery

SUMMARY:
The purpose of this study is compare two different surgical treatments of splenic artery aneurysms: open and laparoscopic approach.

DETAILED DESCRIPTION:
Laparoscopy has not spread into vascular surgery as it has in other surgical branches and still remains in the hands of a minority of surgeons. Splenic artery aneurysm (SAA) is an exception to the rule: an easy-to-reach position and relatively safe control favour the progressive diffusion of laparoscopic techniques.

An increasing number of cases is managed by minimally invasive surgery originating a number of case reports and small series published in recent literature. These papers are unanimous in signalling the feasibility, safety and effectiveness of laparoscopic technique as well as its appreciation by patients -often young females- who harbour the disease. However, perplexities still remain concerning the real potential of laparoscopy in this specific field, in particular considering the spectrum of technical solutions to be performed, the splenectomy rate and the feasibility and results of reconstructive surgery.

The low incidence of the disease justifies the low number of published laparoscopic series enrolling an adequate number of patients and, in particular, the absence of papers comparing open and laparoscopic techniques.

This study reports the first prospective randomized comparison of the different surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Splenic artery aneurysm with diameter greater than 2 cm
* Splenic artery aneurysm with diameter smaller than 2 cm if risk factors for rupture are associated (child bearing age, pregnancy, blister or saccular shape, increasing diameter)

Exclusion Criteria:

* Complex aneurysm involving the celiac trunk
* American Society of Anesthesiologists (ASA) Score > 3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2001-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Overall postoperative morbidity rate | During and after hospital stay, an expected average of 50 months
  According to Dindo-Clavien classification of postoperative complication, we collect in a prospective way and classify all the possible complication by direct clinical evaluation and additional blood sample, imaging or endoscopy if required.

SECONDARY OUTCOMES:
Resumption of oral diet | Partcipants will be followed for the duration of hospital stay, an expected average of one week
  Time between the intervention and patient oral intake without problems
Intra-abdominal surgical drain removal time | Partcipants will be followed for the duration of hospital stay, an expected average of one week
  Time between intervention and removal of surgical drain
Hospital stay length | Partcipants will be followed for the duration of hospital stay, an expected average of one week
  Time between intervention and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Guido AM Tiberio, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Azienda Ospedaliera Spedali Civili di Brescia, Brescia, BS, Italy

REFERENCES:
- [Background] Ha JF, Sieunarine K. Laparoscopic splenic artery aneurysm resection: review of current trends in management. Surg Laparosc Endosc Percutan Tech. 2009 Apr;19(2):e67-70. doi: 10.1097/SLE.0b013e31819bd4e7. PMID 19390269
- [Background] Arca MJ, Gagner M, Heniford BT, Sullivan TM, Beven EG. Splenic artery aneurysms: methods of laparoscopic repair. J Vasc Surg. 1999 Jul;30(1):184-8. doi: 10.1016/s0741-5214(99)70190-4. PMID 10394168
- [Background] Pietrabissa A, Ferrari M, Berchiolli R, Morelli L, Pugliese L, Ferrari V, Mosca F. Laparoscopic treatment of splenic artery aneurysms. J Vasc Surg. 2009 Aug;50(2):275-9. doi: 10.1016/j.jvs.2009.03.015. PMID 19631859
- [Background] Suzuki H, Shimura T, Asao T, Nomoto K, Kanoh K, Tuboi K, Wada S, Kuwano H. Laparoscopic resection of splenic artery aneurysm; a case report. Hepatogastroenterology. 2002 Nov-Dec;49(48):1520-2. PMID 12397723
- [Background] Obuchi T, Sasaki A, Nakajima J, Nitta H, Otsuka K, Wakabayashi G. Laparoscopic surgery for splenic artery aneurysm. Surg Laparosc Endosc Percutan Tech. 2009 Aug;19(4):338-40. doi: 10.1097/SLE.0b013e3181a89206. PMID 19692887
- [Background] Reardon PR, Otah E, Craig ES, Matthews BD, Reardon MJ. Laparoscopic resection of splenic artery aneurysms. Surg Endosc. 2005 Apr;19(4):488-93. doi: 10.1007/s00464-004-8916-8. Epub 2005 Feb 3. PMID 15959711
- [Background] de Csepel J, Quinn T, Gagner M. Laparoscopic exclusion of a splenic artery aneurysm using a lateral approach permits preservation of the spleen. Surg Laparosc Endosc Percutan Tech. 2001 Jun;11(3):221-4. PMID 11444759
- [Background] Sandford RM, Lloyd DM, Ross Naylor A. Laparoscopic ligation of splenic artery aneurysm. Surg Laparosc Endosc Percutan Tech. 2006 Apr;16(2):102-3. doi: 10.1097/00129689-200604000-00010. PMID 16773011
- [Background] Adham M, Blanc P, Douek P, Henri L, Ducerf C, Baulieux J. Laparoscopic resection of a proximal splenic artery aneurysm. Surg Endosc. 2000 Apr;14(4):372. doi: 10.1007/s004640010051. PMID 10854524
- [Background] Meinke AK, Floch NR, Dicorato MP. Laparoscopic options in the treatment of splenic artery aneurysms. Surg Endosc. 2002 Jul;16(7):1107. doi: 10.1007/s00464-002-0003-4. Epub 2002 May 3. PMID 11984676
- [Background] Mastracci TM, Cadeddu M, Colopinto RF, Cina C. A minimally invasive approach to the treatment of aberrant splenic artery aneurysms: a report of two cases. J Vasc Surg. 2005 Jun;41(6):1053-7. doi: 10.1016/j.jvs.2005.01.056. PMID 15944609
- [Background] Holdsworth RJ, Gunn A. Ruptured splenic artery aneurysm in pregnancy. A review. Br J Obstet Gynaecol. 1992 Jul;99(7):595-7. doi: 10.1111/j.1471-0528.1992.tb13828.x. No abstract available. PMID 1525102
- [Background] Ha JF, Phillips M, Faulkner K. Splenic artery aneurysm rupture in pregnancy. Eur J Obstet Gynecol Reprod Biol. 2009 Oct;146(2):133-7. doi: 10.1016/j.ejogrb.2009.05.034. Epub 2009 Jul 10. PMID 19596508
- [Background] Abbas MA, Stone WM, Fowl RJ, Gloviczki P, Oldenburg WA, Pairolero PC, Hallett JW, Bower TC, Panneton JM, Cherry KJ. Splenic artery aneurysms: two decades experience at Mayo clinic. Ann Vasc Surg. 2002 Jul;16(4):442-9. doi: 10.1007/s10016-001-0207-4. Epub 2002 Jul 1. PMID 12089631
- [Background] Jung SI, Joh YG, Um JW, Suh SO, Whang CW, Corbascio M. The Seoul experience of splenic artery aneurysms. Ann Chir Gynaecol. 2001;90(1):10-4. PMID 11336361
- [Background] Pulli R, Innocenti AA, Barbanti E, Dorigo W, Turini F, Gatti M, Pratesi C. Early and long-term results of surgical treatment of splenic artery aneurysms. Am J Surg. 2001 Nov;182(5):520-3. doi: 10.1016/s0002-9610(01)00744-9. PMID 11754862
- [Background] Kokkalera U, Bhende S, Ghellai A. Laparoscopic management of splenic artery aneurysms. J Laparoendosc Adv Surg Tech A. 2006 Dec;16(6):604-8. doi: 10.1089/lap.2006.16.604. PMID 17243878
- [Background] Al-Habbal Y, Christophi C, Muralidharan V. Aneurysms of the splenic artery - a review. Surgeon. 2010 Aug;8(4):223-31. doi: 10.1016/j.surge.2009.11.011. Epub 2010 Mar 12. PMID 20569943
- [Background] Heestand G, Sher L, Lightfoote J, Palmer S, Mateo R, Singh G, Moser J, Selby R, Genyk Y, Jabbour N. Characteristics and management of splenic artery aneurysm in liver transplant candidates and recipients. Am Surg. 2003 Nov;69(11):933-40. PMID 14627251
- [Background] Mattar SG, Lumsden AB. The management of splenic artery aneurysms: experience with 23 cases. Am J Surg. 1995 Jun;169(6):580-4. doi: 10.1016/s0002-9610(99)80225-6. PMID 7771620
- [Background] Moon DB, Lee SG, Hwang S, Kim KH, Ahn CS, Ha TY, Song GW, Jung DH, Ko GY, Sung KB. Characteristics and management of splenic artery aneurysms in adult living donor liver transplant recipients. Liver Transpl. 2009 Nov;15(11):1535-41. doi: 10.1002/lt.21885. PMID 19877249
- [Background] Giulianotti PC, Buchs NC, Coratti A, Sbrana F, Lombardi A, Felicioni L, Bianco FM, Addeo P. Robot-assisted treatment of splenic artery aneurysms. Ann Vasc Surg. 2011 Apr;25(3):377-83. doi: 10.1016/j.avsg.2010.09.014. Epub 2011 Jan 28. PMID 21276711
- [Background] Lee SY, Florica O. Laparoscopic resection of splenic artery aneurysm with preservation of splenic function. Singapore Med J. 2008 Nov;49(11):e303-4. PMID 19037534